CLINICAL TRIAL: NCT03017924
Title: Novel Protection Against Potential Brain, Hearing and Vision Injury During Blast Wave Exposure
Acronym: BLAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-7948
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Q collar (Experimental): Subjects that will wear the Q collar during the breacher training
  Interventions: Device: Q collar
- No collar (No Intervention): Subjects that will not wear the Q collar during the breacher training

INTERVENTIONS:
Device: Q collar — q-collar concussion prevention device
  Arms: Q collar

SUMMARY:
The purpose of the study is to monitor changes in brain structure and function between the pre-training and post-training, in a population of tactical team members wearing the Device and compared to a similar population not wearing the device. Secondly, the purpose is to determine the protection of the device relative to amount and magnitude of sustained head impacts.

DETAILED DESCRIPTION:
This study will investigate the effectiveness of this device in tactical team members exposed to blast waves during tactical training. Subjects participating in this study will be randomly assigned to one of two groups: 1) Device wearing during the tactical training or 2) Non-device wearing during the tactical training. The helmets of all participants will be outfitted with an accelerometer which will measure the magnitude of every concussive blast wave sustained by the subject. Effectiveness of the device will be determined via differences in brain MRI and EEG, vision and hearing testing prior to and following standardized breaching and diversionary device scenario training.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer
* Able to provide written consent

Exclusion Criteria:

* Unable to provide written consent
* History of neurological deficits, previous cerebral infarction, or severe head trauma as indicated through pre-tactical training screening:
* Medical contraindications to restriction of venous outflow via the internal jugular veins (known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Glaucoma (Narrow Angle or Normal Tension)
* Hydrocephalus
* Recent penetrating brain trauma (within 6 months)
* Known carotid hypersensitivity
* Known increased intracranial pressure
* Central vein thrombosis
* Any known airway obstruction
* Any known seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-12; Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Cincinanti Childrens Hospital
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Collar Group: Subjects that will wear the Q collar during the breacher training
  Q collar: q-collar concussion prevention device
- Non-Collar Group: Subjects that will not wear the Q collar during the breacher training
Period: Overall Study
Arm/Group | Collar Group | Non-Collar Group
Started | 12 | 11
Completed | 10 | 8
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Collar Group | Non-Collar Group | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.72 (6.79) | 48.81 (10.37) | 44.27 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 11 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23
Weight [Mean (Standard Deviation); unit: Kg] | 99.10 (17.58) | 93.88 (15.10) | 96.49 (16.34)

OUTCOME MEASURES:

1. Primary Outcome: Blast Explosive Waves Experienced During the Training
Description: The blast explosive waves experienced during the training during the N-back fMRI testing and the rs fMRI testing
Time Frame: single breacher training day
Population: some subjects had head motion during the scan
Measure: Mean (Standard Deviation); unit: number of blasts
Arm/Group | Collar Group | Non-Collar Group
Number analyzed (Participants) | 10 | 9
number of blasts
  Number of blasts N-Back fMRI: number analyzed (Participants) | 9 | 7
  Number of blasts N-Back fMRI | 4.11 (3.37) | 4.29 (2.06)
  Number of blasts rs fMRI | 4.20 (3.19) | 4.0 (2.12)

2. Primary Outcome: Average Peak Pressure Differences Between Groups
Description: between group differences in average peak pressure pre to post in collar versus no collar in both N-back fMRI and rfMRI
Time Frame: Pre-testing appointment occurred 24-48 hours before breacher training and post test appointment occurred 24-48 hours following breached training.
Population: some subjects had head motion
Measure: Mean (Standard Deviation); unit: pounds per square inch
Arm/Group | Q Collar | No Collar
Number analyzed (Participants) | 10 | 9
pounds per square inch
  N-Back fMRI Average peak pressure (psi): number analyzed (Participants) | 9 | 7
  N-Back fMRI Average peak pressure (psi) | 1.67 (0.44) | 1.99 (0.41)
  rs fMRI Average peak pressure (psi) | 1.67 (0.42) | 1.81 (0.53)

3. Secondary Outcome: Between Group Differences in Total Impulse Pre to Post in Collar Versus no Collar
Description: between group differences in total impulse pre to post in collar versus no collar in both the n-back fMRI and the rs fMRI testing conditions
Time Frame: as for outcome 2
Population: All subject data available for this measure - no data lost due to head motion
Measure: Mean (Standard Deviation); unit: units on a scale (psi*ms)
Arm/Group | Collar Group | Non-Collar Group
Number analyzed (Participants) | 10 | 9
units on a scale (psi*ms)
  n-Back fMRI total impulse | 6.58 (4.19) | 7.67 (3.31)
  rs FMRI total impulse | 6.9 (4.08) | 6.95 (3.66)

4. Secondary Outcome: Change in DP-NF Value (Reported in Hz)
Description: pre to post training change in the DP-NF value (the dB difference between the distortion product emission and the noise floor amplitudes) between the collar and no collar groups reported in Hz
Time Frame: as for outcome 2
Population: all subject data available for this analysis
Measure: Mean (Standard Deviation); unit: Change in pre to post Dp (reported in Hz
Arm/Group | Collar Group | Non-Collar Group
Number analyzed (Participants) | 10 | 9
Change in pre to post Dp (reported in Hz
  2000 Hz right | 0.98 (5.10) | 0.64 (3.61)
  2000 Hz Left | 1.64 (6.91) | -0.5 (6.91)
  3000 Hz Right | 5.15 (11.36) | -1.44 (6.47)
  3000 Hz Left | 2.81 (10.28) | -1.29 (10.42)
  4000 Hz right | 5.63 (6.48) | -2.01 (6.85)
  4000 Hz left | 1.54 (7.57) | 2.57 (6.50)
  6000 Hz right | 1.93 (10.40) | -1.29 (8.88)
  6000 Hz left | -1.68 (9.6) | 3.55 (9.24)
  8000 Hz right | 1.43 (6.97) | 1.54 (12.52)
  8000 Hz left | 1.13 (12.21) | 4.23 (9.61)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Collar Group | Non-Collar Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03017924/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03017924/ICF_001.pdf